CLINICAL TRIAL: NCT01202084
Title: A Phase III, Randomized, Open-label, Non-inferiority Study Comparative of Formoterol/Fluticasone Eurofarma 12/250 µg, Foraseq® 12/400 µg and Fluticasone 500 µg in Asthma Patients
Brief Title: A Study Comparative of Formoterol/Fluticasone Foraseq® and Fluticasone in Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 065; CAINAS FF
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2012-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Formoterol/Fluticasone Eurofarma (Experimental): formoterol + fluticasone (12/250 mcg) twice a day per 12 weeks
  Interventions: Drug: Formoterol/Fluticasone
- Foraseq® (Active Comparator): formoterol + budedonide (12/400 mcg) twice a day per 12 weeks
  Interventions: Drug: Foraseq®
- Fluticasone (Active Comparator): fluticasone (500 mcg) twice a day per 12 weeks
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Formoterol/Fluticasone
  Arms: Formoterol/Fluticasone Eurofarma
Drug: Foraseq®
  Arms: Foraseq®
Drug: Fluticasone
  Arms: Fluticasone

SUMMARY:
The primary objective will be to compare the impact of the study formulations on pulmonary function in persistent asthma carriers.

ELIGIBILITY:
Inclusion Criteria:

* Sign the ICF
* Age ≥ 12 years
* Persistent asthma diagnosis, as per the GINA classification (www.ginasthma.com),18 with symptoms for at least 6 months and clinically stable for at least 1 month, with the ACQ-745 test (see Appendix C) ≤ 3.0
* Current use of inhaled corticosteroid (beclomethasone dipropionate dose of up to 1000 µg), associated or not with long-term β2-adrenergic agents and breakthrough medication (salbutamol or equivalent)
* Initial FEV1 of at least 40% of the predicted normal value
* Serum cortisol assessment within normal values.

Exclusion Criteria:

* Use of oral or parenteral corticosteroid within the 3 months prior to study beginning
* Requirement of admission due to asthma within the 3 months prior to study beginning
* Presence of active smoking, defined as the use of cigarette, pipe, cigar or any form of smoking at any amount within the last 3 months
* Presence of severe co-morbidities, such as cardiovascular, renal, liver, neurological, neoplastic, hematological, infectious, dermatological, neurological, psychiatric or chronic respiratory disease other than asthma
* Recent (< 6 months) or predicted participation during this study in other clinical studies involving drugs of any nature or in studies of any form of intervention for treating asthma
* Intolerance or allergy to any of the components of the drugs assessed in the study
* Pregnancy or lactation
* Chronic use of β-blocker medications, per routine oral or intravenous route, or also as ophthalmic solutions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) at final visit. | 12 weeks

SECONDARY OUTCOMES:
Peak expiratory flow (PEF) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- IMA Brasil - Instituto de Pesquisa Clínica e Medicina Avançada, São Paulo, Brazil

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162